CLINICAL TRIAL: NCT06026163
Title: Caffeine for Late Preterm Infants: A Double Blind Randomized Controlled Trial
Brief Title: Caffeine as an Adjuvant Therapy for Late Preterm Infants With Respiratory Distress
Acronym: CAT/LPT
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Fatema Sulaiman Alhazmi, NICU Director, Ministry of Health, Saudi Arabia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-09-M-11
Record Dates: First submitted 2023-08-27; First posted 2023-09-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Prematurity; Respiratory Disease; Ventilator Lung; Newborn
Keywords: caffeine; preterm; newborn; respiratory support
MeSH Terms: conditions — Premature Birth; Respiration Disorders; Bronchopulmonary Dysplasia | interventions — caffeine citrate; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Preparation of caffeine and placebo will be performed by a designated pharmacist who is not part of the study. Parents and investigators will be remained blinded to the administered medications throughout the study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Caffeine citrate group (Experimental): Infants receive either caffeine citrate in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base).
  Interventions: Drug: Caffeine citrate
- Control group (Placebo Comparator): Infants received equivalent volume of saline.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Caffeine citrate — Caffeine citrate in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base)
  Other Names: Intervention group
  Arms: Caffeine citrate group
Other: Placebo — Equivalent volume of saline
  Other Names: Saline
  Arms: Control group

SUMMARY:
Use of caffeine citrate in late-preterm infants with respiratory distress is questionable. Oliphant and colleagues found in a recently published study that caffeine therapy use in late-preterm infants at a loading dose of 20 and 40 mg/kg and maintenance dose of 10 and 20 mg/kg/day reduces the incidence of intermittent hypoxia events by 61 and 67% respectively.

The investigators hypothesized that caffeine will improve respiratory drive, prevent apnea, shorten the hospital stay and improve arousal state in late preterm infants.

The investigators aim to study the effect of caffeine citrate on late preterm babies as regard duration of respiratory support, duration of hospital stay, respiratory morbidity, incidence and frequency of apnea.

DETAILED DESCRIPTION:
late preterm infants will be randomized in a blinded manner to receive either caffeine in loading dose 20 mg/kg (equivalent for 10 mg/kg caffeine base) and maintenance dose 10 mg/kg/day (equivalent for 5 mg/kg caffeine base) in Caffeine treatment group, or equivalent volume of saline in the placebo group. Caffeine will be continued until infants get off all forms of respiratory support.

Preparation of caffeine and placebo will be performed by a designated pharmacist who is not part of the study. Parents and investigators will be remained blinded to the administered medications throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants at gestational age 34 0/7 through 36 6/7
* Presented with respiratory distress
* Require respiratory support in the form of any of the following :

A) Invasive mechanical ventilation, B) Non-invasive positive pressure ventilation, C) Nasal cannula with FIO2 requirement over 50% to keep pre-ductal saturation between 90-95%.

Exclusion Criteria:

1 - Late preterm admitted for non-respiratory etiologies 2- Late preterm infants requiring nasal cannula on less than 50% FIO2 by 4 hours of age as they are less likely to require respiratory support for a long time.

3- Newborn infants with congenital malformations and chromosomal anomalies. 4- Infants with echocardiographic evidence of PPHN requiring medical intervention.

5- Late preterm with history of maternal substance abuse

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Duration of respiratory support | 28 days
  cumulative duration of mechanical ventilation, non-invasive positive pressure ventilation and nasal cannula therapy (days)

SECONDARY OUTCOMES:
Episodes of apnea | 28 gays
  the cessation of breathing for more than 20 seconds or cessation of breathing for accompanied by bradycardia or desaturation
Failure of extubation | 28 days
  need of re-intubation within 72 h of extubation from mechanical ventilation
Duration of caffeine | 28 days
  Days of caffeine treatment
Length of hospital stay | 28 days
  days of hospital admission
Time to full enteral and oral feeding | 28 days
  days to reach full enteral feeds
Adverse effects of caffeine use | 28 days
  Tachycardia, irritability, feeding intolerance, hypertension
Caffeine withhold | 28 days
  Caffeine withhold for suspected side effects
Weight gain per day | 28 days
  Weight gain per day (gram)
Mortality | 28 days
  Death before hospital discharge
Readmission rate | 28 days
  Readmission to the hospital with respiratory related symptoms within 48 hours of hospital discharge
Days of apnea | 28 days
  Days of apnea

CONTACTS AND LOCATIONS:
Overall Officials: Nehad Nasef, Principal Investigator — Neonatology Consultant
Locations (2):
- Saudi Arabia (2):
  - King Salman Bin Abdulaziz Medical City, Madinah, Medina Region
  - King Salman Bin Abdulaziz Medical City, Madinah

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers for research and scientific purposes (i.e conduction of meta-analysis or systematic review). Data or samples shared will be coded, with no protected health information included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol
Time Frame: Data requests can be submitted starting 3 months after article publication and the data will be made accessible for up to 12 months. Extensions will be considered on a case-by-case basis."
Access Criteria: Access to raw data (no protected health information) can be requested by qualified researchers for scientific purposes, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA)

REFERENCES:
- [Background] Davis PG, Schmidt B, Roberts RS, Doyle LW, Asztalos E, Haslam R, Sinha S, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine for Apnea of Prematurity trial: benefits may vary in subgroups. J Pediatr. 2010 Mar;156(3):382-7. doi: 10.1016/j.jpeds.2009.09.069. Epub 2009 Nov 18. PMID 19926098
- [Background] Eichenwald EC; Committee on Fetus and Newborn, American Academy of Pediatrics. Apnea of Prematurity. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3757. Epub 2015 Dec 1. PMID 26628729